CLINICAL TRIAL: NCT06693544
Title: Comparing Intracellular Anabolic Capacity and Food-derived Amino Acid Bioavailability of Peanut and Dairy Protein in Healthy Non-frail Older Adults at Risk for (Pre)Frailty
Brief Title: Peanut Sip Feeding Protocol
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Professor, Texas A&M University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 98-Peanut
Record Dates: First submitted 2024-10-11; First posted 2024-11-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Protein Metabolism
Keywords: Prandial; Plant protein; Animal protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy male older adults (Experimental)
  Interventions: Dietary Supplement: Peanut protein
- Healthy female older adults (Experimental)
  Interventions: Dietary Supplement: Peanut protein

INTERVENTIONS:
Dietary Supplement: Peanut protein — Commercially available plant-based protein powders

SUMMARY:
Peanuts are considered a functional food and regular consumption is associated with positive health effects. Protein is the second most common nutrient in peanuts after fat. The protein digestibility of peanuts is similar to that of animal protein, and the limiting amino acids in peanuts vary based on the study and are suggested to be lysine, methionine, or threonine. Defining the reduced responsiveness of various dietary proteins to induce anabolism in older adults is critical for preventing and attenuating physical and cognitive health decline.

DETAILED DESCRIPTION:
The study will be conducted in healthy, non-frail older adults, stratified into different age categories. A sip feeding model will be used as it is a good model to establish the anabolic capacity of meals.Our research objective is to examine whether differences exist in the anabolic response and bioavailability of amino acids coming from peanut-based protein as compared to animal-based protein in older adults at risk for (pre-)frailty, known to contribute to poor muscle and brain health. The study will take place at the research facility of the Center for Translational Research on Aging and Longevity (CTRAL), Texas A&M University located in the Human Clinical Research Building ) affiliated with Texas A&M University. The study involves 1 screening visit of approx. 3 hours, and 4 study days. Some study procedures (e.g., body composition, skeletal muscle function, questionnaires) may be skipped if completed within the past 3 months at CTRAL. All data will be recorded in Case Report Form and stored in the Texas A&M REDCap System. Subjects will be asked to arrive in the fasted state on all study days. Fasting prior to screening is not required. On the screening day, body weight, height, and body composition by Dual-energy X-ray absorptiometry (DXA) will be measured. In addition, The Six-Minute Walk Test (6MWT) and skeletal muscle function tests will be assessed at the end of each screening visit. Each study visit will begin with vital signs. Before administration of the feeding or the tracer solution, baseline blood will be collected for measurement of the natural enrichment of metabolites. After the baseline sample is collected, feeding will begin and will be followed by tracers of several compounds that may be administered by IV pulse. Participants will receive the liquid nutritional supplement as sip feeds every 20 minutes for 5 hours. The liquid nutrition supplements will contain 45g of peanut protein (plant based). Comparison of results from meals taken while enrolled in NCTNCT06628349 will be performed. Participants will have the option of adding sugar free (SF) vanilla syrup, SF caramel syrup, or SF chocolate syrup to their meals.

ELIGIBILITY:
Inclusion criteria:

* Previous completion of IRB2023-0549: Prandial Metabolic Phenotyping in Sarcopenic Older Adults Comparing Plant Based and Whey Based Protein (NCT06628349)
* Age 65-80 years old
* Stable body-weight (less than ±5% in the previous 6 months)
* Ability to walk, sit down, and stand up (independently or with walking assistance device)
* Willingness to lay supine in bed for up to 6 hours
* Willingness and ability to comply with the protocol

Exclusion criteria

* Established diagnosis and active treatment of chronic disease: Insulin dependent diabetes mellitus, active malignancy, heart disease, kidney disease, liver disease, HIV/AIDS, Asthma (moderate to severe), Hep (A,B, or C)
* History of untreated metabolic disease including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Active dependence of alcohol or drugs
* Use of short course of oral corticosteroids within 4 weeks preceding study day
* Current use of long-term oral corticosteroids
* Use of protein or amino acids containing nutritional supplements within 5 days of the first study day
* Planned elective surgery requiring 2 or more days of hospitalization during the entire study
* (Possible) pregnancy
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject
* Already enrolled in another clinical trial
* Any condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* Known allergy to any of the components of the feeding (i.e., peanut)
* Experienced issue with intake of peanut or peanut products within the previous year
* Established daily diet of vegetarian / vegan composition

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Protein synthesis capacity of plant-based in older adults without sarcopenia measured by the use of stable isotope tracers | 2 weeks
  A novel stable isotope technique will be used to assess simultaneously the anabolic response and whole-body production rates of protein synthesis when taking oral nutrition in sarcopenic older participants. The samples will be stored in laboratory freezers and the amino acid isotope enrichments and concentrations analyzed by Liquid Chromatography with tandem mass spectrometry (LC-MS/MS). The researchers will then conduct LC-MS/MS analysis, peak integration, calculation of amino acid concentrations and whole body productions from raw data, and use the results for preparation of papers for presentation, publication, and final reports. The researchers main hypothesis is that plant-based protein induces less protein anabolism, due to lower whole body production of essential amino acids (EAA) and higher production of non-essential amino acids (NEAA).

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University - CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared upon request for up to 6 years beyond completion of the trial based on methods/proposals approved by both parties' institutional review committees. Individual participant data that underlie the results of the trial may be shared after de-identification (text, tables, figures, and appendices). Additional documents available per request include: study protocol, statistical analysis plan, and informed consent. Requests should be directed to Dr. Marielle Engelen (mpkj.engelen@ctral.org).

DOCUMENTS (1):
  • Informed Consent Form (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT06693544/ICF_000.pdf